CLINICAL TRIAL: NCT07105072
Title: Outcomes of Vitrectomy Versus Suprachoroidal Steroid Injection in Cases of Presumed-trematode Induced Granulomatous Intermediate Uveitis
Brief Title: Vitrectomy Versus Suprachoroidal Steroid in Trematodal Granulomatous Uveitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ekram Mohamed Rabie, Assisstant Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Intermediate uveitis
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Trematode Induced Granulomatous Uveitis
Keywords: Trematode-Uveitis-Steroid-Vitrectomy
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitrectomy arm (Active Comparator): Pars Plana vitrectomy and debulking of ciliary body granuloma
  Interventions: Procedure: Vitrectomy
- Suprachoroidal steroid injection (Active Comparator): Suprachoroida steroid injection of triamcinolone acetonide for ciliary body granuloma.
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — vtrectomy is a surgical procedure to remove vitreous humor and can be used in case of viritis and as a debulking procedure for ciliary body granuloma.

SUMMARY:
Presumed trematode-induced granulomatous intermediate uveitis (PTIGIU) presents with vitritis and complicated cataract (active stage) which, if left untreated, progresses to tractional retinal detachment (TRD) from the vitreoretinal traction (cicatricial stage) and eventually cilliary body shut down and atrophia bulbi Accordingly, timely diagnosis of such patients during the active stage is essential for early proper management to avoid complications that might eventually result in blindness.

Many treatment modalities for the treatment of AC granulomas were reported, including various combinations of topical corticosteroids, systemic antiparasitic treatment, peribulbar anterior subtenon steroids injections and surgical granuloma excision. Resistant cases may be treated with oral prednisone starting at a daily dose of 1 mg/kg which is gradually tapered over 3-6 weeks . Therefore, many cases may develop steroid-related complications such as cataracts and glaucoma.

This study aims at comparing 6-month visual outcomes and complications after vitrectomy versus suprachoroidal triamcinolone acetonide (SCTA) injection in patient presented with cilliary body granuloma in Presumed trematode-induced granulomatous intermediate uveitis (PTIGIU).

DETAILED DESCRIPTION:
Microbial infections such as tuberculosis, toxocariasis, and toxoplasmosis can induce granulomatous uveitis in children. Also, it might be induced by non-infectious causes such as sarcoidosis, sympathetic ophthalmia, or Vogt-Koyanagi-Harada disease. Also, parasitic infestation of the eye can produce significant granulomatous uveitis with subsequent complications. Presumed trematode-induced uveitis most frequently observed in children who swim in nearby freshwater canals harboring trematode-infected snail. The term "presumed" is used to describe this type of uveitis as fragments and genetic material of the parasites could be isolated from only some of the surgically removed granulomas without signs of systemic parasitic disease. The hallmark of trematode-induced granulomatous inflammation is one or more pearl-like nodules almost always seen in the inferior quadrant of the anterior chamber (AC), which has been documented in Egypt and India. Sometimes, intermediate uveitis with snow banking and cilliary body granuloma, lens granuloma, iris granulomas and posterior uveitis could be the presenting feature of this disease. Less frequently, subconjunctival lesions or corneal lesions can also occur.

Ocular inflammation may be secondary to the reaction of the immune system of the host against the parasite or its toxic products.

Procerovum varium, a trematode, was identified as the causative agent responsible for AC granuloma in children in South India. Schistosomiasis, also known as bilharziasis, is an endemic disease caused by trematodes of the Schistosoma genus in Egypt. Relatively rare ocular involvement has been attributed to Bilharziasis, mainly in the form of granuloma reaction induced by the ova or adult worms in different ocular tissues. Schistosoma mansoni was also observed and isolated from the AC angle. The cercariae (infective stage) of the trematode can reach maturity and lay ova directly in the veins of the richly vascularized conjunctiva, which subsequently leads to the development of sub-conjunctival granuloma. In some cases, cercariae can penetrate limbal structures and gain access to the anterior chamber leading to the development of AC granuloma. This has been considered the most accepted theory that explains how the ova of the trematode or adult worms reach the eye.Case reports have traced the life cycle of the parasite Procerovum varium in patients with trematode granuloma. It is a trematode found in the conjunctival sac of the birds. When these birds come into contact with the water bodies, the adult worms from the conjunctival sac can release eggs into these reservoirs. These eggs can then hatch into miracidia. When miracidia infect the intermediate host, the snails, the miracidia mature to become cercariae. These cercariae to complete their life cycle have to reach the birds again. Humans are accidental hosts in this cycle. Children are affected when they come in contact with the water infested with the cercariae. The parasite directly enters the eyes penetrating the ocular tissues.

The ocular manifestations can be caused by either direct trauma from the parasite or secondary to the toxic products released by the organisms. There are multiple theories as to how the trematode reaches the ocular tissue. Alternatively, the trematode ova can also reach the ocular tissue from systemic circulation after it matures to cercariae. They lay eggs in the highly vascularized conjunctiva, deep episcleral plexus, limbus and anterior chamber.

Whatever be the mode of entry of these parasites, the final pathology is that the released ova cause inflammation which leads to a granulomatous reaction in the ocular tissue. The granuloma is found to have teguments or internal fragments of parasites in the centre of the lesion surrounded by neutrophils, eosinophils. mononuclear cells, lymphocytes, macrophages, multinucleated giant cells and fibroblasts. Splendore-Hoeppli phenomenon is described in the histopathological evaluation of a few granulomas in the study by Rathinam et al. and others. Splendore-Hoeppli phenomenon is characterized by the presence of radiating intensely eosinophilic material around the parasite. Finally, when the inflammation settles down, there is deposition of collagen in the places of granuloma.

Clinical course In geographical areas, where the water reservoirs are infested with the parasite, the patients usually children can present with itching, erythema after a bath in the pond. Few of them develop swelling of the buccal and genital mucosa. These systemic occurrences are self-limiting and recalled by the patient only while questioning during ocular evaluation.

The ocular presentation occurs when the organism penetrates the ocular tissues like the episcleral or anterior chamber, sometimes even the lid structures. These patients may present with anterior chamber granuloma with or without granulomatous uveitis. Few may have both subconjunctival and anterior chamber granuloma. The disease is usually unilateral, but in rare instances can be bilateral. Anterior chamber granuloma can be single or multiple. Mostly these lesions are at the angle with or without granulomatous reaction associated with the lesion.

Symptoms Usually, these are young boys who presented with granuloma to us, as the social norms do not allow girls to take baths in open water reservoirs in the village communities. The chance of infection is less in children younger than 4 years, as they do not tend to take baths in water bodies for longer duration. These boys presented to the ophthalmologist with pain, redness or a white mass seen in the eye. Rarely a child can present with lid swelling. Usually, there will be a preceding history of taking baths in water bodies for a longer duration before presenting with such ocular inflammation. On proper reviewing, a history of similar presentations can be elicited in other children or siblings who have taken part in similar activities in their region.

Signs This disease can be unilateral or bilateral. The common presentation can be subconjunctival granuloma, anterior chamber granuloma with granulomatous keratic precipitates and grade 1 to 2 + cells. These lesions are white and well-circumscribed and can be sub mm to 2.5 mm and larger in diameter. They can be single or multiple. Cataracts can be seen in few children during the course of the disease or when they present very late. The retro corneal membrane is seen in few patients. Lid swelling mimicking chalazia can be the presenting sign and can be misdiagnosed if proper history-taking and knowledge towards the geographical belt is not present.Cataracts and glaucoma are late complications in few of these children due to chronic inflammation.

Recently few cases were reported with intermediate uveitis associated with ciliary body granuloma. However, these cases are not proven by molecular diagnostics.The author has relied only on temporal association with exposure to water bodies.

Prevention In conclusion, when there is a clustering of similar cases, with no appropriate aetiology, endemic infection has to be suspected. We can understand establishing an aetiology in such cases is a long journey and this article has tried to trace the history of the trematode granuloma from the point of origin (snails in river bed) to the point of identification (PCR/molecular diagnostics). The primary treating physician should have a knowledge of the locally occurring diseases or else these children may be treated as tuberculous uveitis. Again, the local bodies should be educated about these diseases to prevent further occurrences. Knowledge, attitude and practice towards the disease have to be improved both among the general public and the doctor population to reduce the incidence.

Suprachoroidal steroid injection Suprachoroidal steroid injections, such as triamcinolone acetonide, are being explored as a treatment option for presumed-trematode induced granulomatous intermediate uveitis, particularly when conventional treatments are insufficient. These injections aim to deliver medication directly to the posterior segment of the eye, potentially improving efficacy and reducing side effects associated with other steroid delivery methods. [52] • Presumed-Trematode Induced Granulomatous Intermediate Uveitis [53]: This refers to inflammation of the middle layer of the eye (uvea) that is thought to be caused by parasitic trematode infections, specifically the formation of granulomas (small masses of immune cells).

• Intermediate Uveitis: This type of uveitis affects the vitreous (the gel-like substance in the eye) and the peripheral retina.

• Suprachoroidal Injection: This involves injecting medication into the suprachoroidal space, a potential space between the sclera (outermost layer of the eye) and the choroid (the vascular layer).

• Targeted Delivery: Suprachoroidal injections allow for higher drug concentrations in the posterior segment of the eye compared to other methods, potentially improving treatment effectiveness.

• Reduced Side Effects: By delivering medication directly to the site of inflammation, suprachoroidal injections may reduce the risk of systemic side effects associated with oral corticosteroids and reduce the risk of steroid-related complications in the eye, such as cataracts and elevated intraocular pressure.

• Alternative to Conventional Treatments: When conventional treatments like topical or oral corticosteroids are not sufficient or cause unacceptable side effects, suprachoroidal injections offer a potential alternative.

Clinical Evidence and Research:

• Positive Results: Studies have shown that suprachoroidal triamcinolone acetonide injections can improve visual acuity and reduce macular edema in patients with uveitis.

• Safety Profile: While some side effects like eye pain or elevated intraocular pressure can occur, the overall safety profile of suprachoroidal injections appears favorable, especially in comparison to other corticosteroid administration methods.

Further research is being conducted to evaluate the long-term efficacy and safety of suprachoroidal injections in various types of uveitis, including those presumed to be caused by trematodes.

In the context of presumed-trematode induced granulomatous intermediate uveitis, suprachoroidal injections are being investigated as a promising treatment option that may offer improved efficacy and a better safety profile compared to other methods, particularly when conventional treatments are not effective or cause significant side effects.

ELIGIBILITY:
Inclusion Criteria:

* Children with history of fresh canal water exposure prior to the onset of uveitis.
* Intermediate uveitis with CB granuloma detected by ultrasound biomicroscopy (UBM).
* Absence of clinical signs or work-up suggestive of any other cause of granulomatous intermediate uveitis.
* Failure of medical treatment was defined as persistent or recurrent anterior (flare and cells >+1) and/or posterior segment inflammation (>Grade I vitritis) following oral steroids for 8-12 weeks as reported in previous literature.

Exclusion Criteria:

* Co-existing ocular pathology that could influence the final visual acuity (VA).
* known cause of granulomatous uveitis other than trematodal such as(Tuberculosis, sarcoidosis, Syphilis, toxoplasmosis, toxocariasis, Juvenile idiopathic arthritis)
* Evidence of ocular trauma
* previous ocular surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Size | From enrollment to the end of treatment at 6 months
  Size of ciliary body granuloma by UBM
Size of ciliary body granuloma | six months follow up
  Using Ultrasound biomicroscopy for measuring ciliary body granuloma

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Minia university, Minya, Egypt

REFERENCES:
- [Result] Amin RH, Abdullatif AM. Management of presumed trematode-induced granulomatous intermediate uveitis. Eye (Lond). 2023 Aug;37(11):2299-2304. doi: 10.1038/s41433-022-02336-4. Epub 2022 Dec 7. PMID 36477731